CLINICAL TRIAL: NCT02346474
Title: Cross Calibration of Two Dual Energy Densitometers and Comparison of Regional Adipose Tissue Measurements by iDXA and MRI.
Status: Completed | Type: Observational
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999915054; 15-DK-N054
Record Dates: First submitted 2015-01-24; First posted 2015-01-27 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Obesity
Keywords: Subcutaneous Fat; Visceral Fat
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- It is important for doctors to know how much fat a person has in his or her body. Machines called DXAs measure how much fat mass and fat-free mass a person has. Researchers in this study have a new DXA machine, and they want to know if it measures body fat as well as the old machine. They also want to see how body fat readings from the new DXA compare to readings from a magnetic resonance imaging (MRI) scan.

Objectives:

- To see if two DXA machines give the same results when measuring body fat. Also, to know whether the DXA and MRI give the same results in measuring visceral and subcutaneous fat.

Eligibility:

- People 18 years and older who weigh less than 350 pounds.

Design:

* Participants will be screened with a medical history and physical exam. Women will have a pregnancy test. Researchers will make sure participants are able to have an MRI if they volunteered to.
* Participants will have their body fat measured by each DXA scanner. They will lie quietly on a padded table while being scanned. The scan uses X-rays to take pictures of the body. Both scans will be done on the same morning and will take 10-15 minutes on both machines.
* Some participants also will have their body fat measured with MRI. They will lie in a long, tube-shaped scanner. The machine uses strong magnetic fields and radio waves to take pictures of internal organs. Participants will sign an additional consent form for this procedure.

DETAILED DESCRIPTION:
Our Research unit (NIDDK) recently acquired a new x-ray unit (the General Electric (GE) Lunar iDXA) for measurement of body composition (how much fat someone has as a percent of their weight). This machine provides clearer and crisper images. The unit also has a larger table to allow patients up to 450 lbs (204 kg) to be scanned. The larger table allows for easier positioning of tall and heavy patients. We would like to use this new machine in the future but want to see whether our current DXA unit (the Lunar Prodigy Densitometer by GE) and the Lunar iDXA Densitometer (GE) measure the same percentage of a person s body fat. If there are measurement differences between the two machines, we will develop a way to convert the new results to more closely match the results from the current DXA unit. Thus, in this study, we will be asking volunteers to undergo scanning for measurement of body fat on both machines on the same day.

Fat within the belly which is around organs (called visceral fat or VAT) is linked to more bad health outcomes than fat which is just underneath the skin (called subcutanoues fat or SAT). Along with standardizing the DXA - body composition measurement results we would like to compare VAT and SAT estimates from iDXA with values obtained by MRI. The precise MRI measurements completely avoid radiation exposure for the volunteers but are far more time consuming. Knowing that the results of iDXA match up with or correlate with the MRI results would allow us to use iDXA measurements to estimate visceral and subcutaneous adipose tissue depots in ongoing and the future studies.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Age range: greater than or equal to 18 years old
  2. Individuals will be recruited to represent a broad range of BMI such that approximately equal numbers of men and women in BMI groups of < 25 kg/m(2), greater than or equal to 25 kg/m(2)-<30 kg/m(2), and greater than or equal to 30kg/m(2) are represented.
  3. NIH employees will be allowed to participate

EXCLUSION CRITERIA:

1. Individuals who, based on their radiation history and by our local radiation exposure reports, would exceed the safety limits imposed by current Phoenix Radiation Safety Committee radiation safety guidelines.
2. Pregnant females, due to exposure to research related radiation in this study
3. Presence of a pacemaker or other implantable devices/shrapnel which may interfere with the MRI scan.
4. Central nervous system disease ( such as cerebrovascular accidents, dementia, and neurodegenerative disorders) which preclude individuals from being able to provide informed consent.
5. Current or past history of: bipolar disorder, schizophrenia or presence of psychotic symptoms, bulimia nervosa or anorexia nervosa, or current major depressive disorder which preclude individuals from being able to provide informed consent.
6. Weight > 350 pounds (limit of currently used DXA scan)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01-24 (Actual); Primary Completion 2016-07-28 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Comparison of body fat measurements | 1 year

SECONDARY OUTCOMES:
Comparison of DXA and MRI visceral fat | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Krakoff, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

REFERENCES:
- [Derived] Reinhardt M, Piaggi P, DeMers B, Trinidad C, Krakoff J. Cross calibration of two dual-energy X-ray densitometers and comparison of visceral adipose tissue measurements by iDXA and MRI. Obesity (Silver Spring). 2017 Feb;25(2):332-337. doi: 10.1002/oby.21722. Epub 2016 Dec 21. PMID 28000375